CLINICAL TRIAL: NCT02769988
Title: Focus Group Evaluation of Educational Impact of the NLM / National Area Health Education Center Organization (NAO) Project-SHARE Based Teen Health Information Literacy Curriculum
Brief Title: Educational Impact of the NLM/National Area Health Education Center Organization (NAO) Project-SHARE Based Teen Health Information Literacy Curriculum
Status: Completed | Type: Observational
Sponsor: National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916100; 16-LM-N100
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2018-06-26

CONDITIONS: Healthy Volunteers Only
Keywords: Adolescents; Health Information Literacy; Health Education
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Project SHARE

SUMMARY:
Background:

The Teen Health Information Literacy Project is an after-school program for high school students. It gives them skills to access valid and reliable health data. It also aims to grow young health advocates. Researchers want to find out more about the impact the program has had on students. They want to use this feedback to improve the program.

Objective:

To gain feedback about the Teen Health Information Literacy Project.

Eligibility:

Young people who participated in the Teen Health Information Literacy Project. The project was run by Area Health Education Centers (AHECs) and sponsored by the National Library of Medicine (NLM).

Design:

The study will be explained to students during a program session. They will take consent forms home to their parents.

Participants will split into 6 focus groups. Each one will be conducted at an AHEC project site.

The focus group will be a 90-minute discussion between participants and an evaluator from the NLM. The evaluator will be present either in person or by video conference.

The evaluator will ask participants questions, which may include the following. What did they like and dislike about the program? Why did they decide to participate? What have they learned? Would they recommend this program to another student? How has the program affected their interest in health-related careers?

The discussion will be audio-recorded. The evaluator will use an automated tool to convert recordings into text. After that, she will destroy the audio.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the impact of the National Library of Medicine (NLM)/ National Area Health Education Center Organization (NAO) Teen Health Information Literacy Curriculum (based on an earlier Project SHARE curriculum) on the participants : understanding of health disparities in their communities; leadership, health advocacy, and communication skills; sense of self and connectedness with the community; and interest in health-related careers. Study population: The study population consists of program participants at the five participating sites, which include local AHEC chapters of Boston, Brooklyn-Queens-Long Island, Colorado, Eastern Connecticut, and Montana. The program participants are middle and high school students, ranging in ages from 13 to 18 years old. All participants will be invited to participate. Design: The study will involve moderated focus groups at each participating site. Outcome measures: participants understanding of health disparities in their communities; leadership, health advocacy, and communication skills; sense of self and connectedness with the community; and interest in health-related careers.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participation in the NLM / NAO Teen Health Information Literacy Project

EXCLUSION CRITERIA:

-NA

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 127 (Actual)
Dates: Start 2016-05-11; Primary Completion 2016-10-05 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Participant's understanding of health disparities in their communities; leadership, health advocacy, and communication skills; sense of self and connectedness with the community; and interest in health-related careers | End of Program

CONTACTS AND LOCATIONS:
Overall Officials: Alla Keselman, Ph.D., Principal Investigator — National Library of Medicine (NLM)
Locations (6):
- United States (6):
  - SW Colorado AHEC, Durango, Colorado
  - Centennial AHEC, Greeley, Colorado
  - Eastern CT AHEC, New London, Connecticut
  - Boston AHEC, Boston, Massachusetts
  - Montana AHEC, Bozeman, Montana
  - Bqli Ahec, Queens, New York